CLINICAL TRIAL: NCT01611558
Title: A Phase II Safety and Efficacy Study of Ipilimumab Monotherapy in Recurrent Platinum Sensitive Ovarian Cancer Subjects
Brief Title: Phase II Study of Ipilimumab Monotherapy in Recurrent Platinum-sensitive Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA184-201
Record Dates: First submitted 2012-05-25; First posted 2012-06-05 (Estimated); Results first posted 2016-04-19 (Estimated); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Platinum-sensitive Ovarian Cancer, Second-line, Third-line, or Fourth-line
MeSH Terms: interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm: Ipilimumab, 10 mg/kg (Experimental): Participants received 10 mg/kg of ipilimumab administered intravenously once every 3 weeks for 4 doses (Induction Phase). Then, once every 12 weeks (Maintenance Phase), until disease progression or unacceptable toxicity occurs.
  Interventions: Biological: Ipilimumab

INTERVENTIONS:
Biological: Ipilimumab
  Other Names: Yervoy; BMS-734016

SUMMARY:
To assess the incidence of drug-related adverse events of Grade 3 or higher and the overall response associated with ipilimumab treatment

DETAILED DESCRIPTION:
Condition: Ovarian Cancer, Second line, Third line, or Fourth line

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Key Inclusion Criteria

* Ovarian cancer that is not refractory or resistant to platinum-based therapy (refactory=progression while receiving any previous platinum regimen; resistant=progression within 6 months of any previous platinum regimen)
* Recipients of platinum/taxane-based chemotherapy as frontline regimen for ovarian cancer
* An Eastern Cooperative Oncology Group performance status ≤1
* Up to 4 prior lines of therapy for ovarian cancer
* Two groups are eligible:

Group 1. Women who have not met the criteria for progressive disease following their most recent chemotherapeutic regimen were required to have:

* Demonstrated partial response or stable disease following the most recent chemotherapy regimen
* Evaluable or measurable disease, detected by baseline computed tomography (CT) or magnetic resonance imaging (MRI) scan
* Received the last dose of their most recent chemotherapeutic regimen for ovarian cancer within 4 to 12 weeks of the first administration of ipilimumab Group 2: Women with disease progression while receiving or following the last dose of the most recent chemotherapeutic regimen were required to have:
* Measurable disease on a CT or MRI scan performed within 28 days of first dose of ipilimumab.
* Received the last dose of their most recent chemotherapeutic regimen for ovarian cancer at least 4 weeks prior to the first administration of ipilimumab.

Key Exclusion Criteria

* Histologic diagnosis of borderline, low malignant potential epithelial carcinoma
* For Group 1, women with complete response on the most recent ovarian carcinomatherapy
* Presence of known brain metastases
* Second malignancy active within the past 5 years, with the exception of locally curable cancers that have no need for subsequent therapy
* Documented history of severe autoimmune or immune-mediated symptomatic disease requiring prolonged systemic immunosuppressive treatment
* History of motor neuropathy considered to be of autoimmune origin or the of grade 2 or higher peripheral neuropathy
* History of toxic epidermal necrolysis
* Prior therapies with immunosuppressive agents within the last 2 years (excluding low-dose corticosteroids) and prior therapies with cytotoxic drugs within 4 weeks
* Chronic use of systemic immunosuppressive drugs, ongoing use of immunotherapy or biologic therapy for the treatment of cancer, or prior use of ipilimumab or any immune-stimulating agent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-08-21 (Actual); Primary Completion 2014-11-03 (Actual); Study Completion 2019-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (17):
- United States (17):
  - Yale University School Of Medicine, New Haven, Connecticut
  - AdventHealth Cancer Institute, Orlando, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute., Atlanta, Georgia
  - Georgia Regents University, Augusta, Georgia
  - Dr. Sudarshan K. Sharma, Ltd., Hinsdale, Illinois
  - Indiana University Health Melvin And Bren Simon Cancer Center, Indianapolis, Indiana
  - Women'S Cancer Care, Covington, Louisiana
  - Dana Farber Cancer Institute., Boston, Massachusetts
  - Memorial Sloan Kettering Nassau, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - The Charlotte-Mecklenburg Hospital Authority, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - Peggy and Charles Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute, LLC, Tulsa, Oklahoma
  - Magee-Womens Hospital Of Upmc, Pittsburgh, Pennsylvania

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 40 participants enrolled and treated
Groups:
- Ipilimumab, 10 mg/kg: Participants received 10 mg/kg of ipilimumab administered intravenously once every 3 weeks for 4 doses (Induction Phase). Then, once every 12 weeks (Maintenance Phase), until disease progression or unacceptable toxicity occurs.
Period: Induction Phase
Arm/Group | Ipilimumab, 10 mg/kg
Started | 40
Completed | 2
Not Completed | 38
Not completed — Study drug toxicity | 15
Not completed — Disease progression | 18
Not completed — Heart arrest,urosepsis,respiratory fail | 1
Not completed — Adverse event unrelated to study drug | 3
Not completed — Death | 1
Period: Maintenance Phase
Arm/Group | Ipilimumab, 10 mg/kg
Started | 2
Completed | 0
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Elevated Uric acid | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug
Groups:
- Ipilimumab,10 mg/kg: Participants received 10 mg/kg of ipilimumab administered intravenously once every 3 weeks for 4 doses (Induction Phase). Then, once every 12 weeks (Maintenance Phase), until disease progression or unacceptable toxicity occurs.
Arm/Group | Ipilimumab,10 mg/kg
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: Years] | 61.5 [42.0 to 74.0]
Age, Customized [Count of Participants; unit: Participants]
  Younger than 65 years | 28
  65 years and older | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 35
  Black or African American | 2
  Asian | 2
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Drug-related Adverse Events (AEs) of Grade 3 or Higher
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. Treatment-related=having certain, probable, possible, or missing relationship to study drug. Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4=Potentially Life-threatening or disabling.
Time Frame: Day 1, first dose, to within 90 days of last dose in Induction Phase
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Ipilimumab, 10 mg/kg
Number analyzed (Participants) | 40
Participants | 20

2. Secondary Outcome: Best Overall Response Rate (BORR)
Description: BORR is defined as the percentage of participants who received treatment and, at any time during the study, had a best response of complete response or partial response, as confirmed by Response Evaluation Criteria in Solid Tumors (RECIST) or Rustin criteria for patients with cancer antigen 125 (CA125) levels elevated to twice the upper limit of normal at baseline, divided by the total number of evaluable participants in the arm.
Time Frame: From first dose of study drug to unacceptable toxicity or progressive disease (to a maximum of 3 years)
Population: All participants who received study drug. n=number of evaluable participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ipilimumab,10 mg/kg
Number analyzed (Participants) | 40
Percentage of participants | 15.0 [5.7 to 29.8]

3. Secondary Outcome: Number of Participants Who Died and With Serious Adverse Events (SAEs), Drug-related SAEs, Drug-related AEs, AEs Leading to Discontinuation, and Drug-related AEs Leading to Discontinuation
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. Treatment-related=having certain, probable, possible, or missing relationship to study drug.
Time Frame: From first dose to within 90 days of last study dose
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Ipilimumab,10 mg/kg
Number analyzed (Participants) | 40
Participants
  Deaths | 35
  SAEs(induction phase) | 26
  Drug-related SAEs | 16
  Drug-related AEs | 38
  AEs leading to discontinuation | 16

ADVERSE EVENTS:
Time Frame: On or after Day 1 of study treatment and no later than 90 days following the last day of study treatment ( Up to 5 years).
Arm/Group | 10 mg/kg Ipilimumab
All-Cause Mortality (participants affected / at risk) | 35/40
Serious Adverse Events (participants affected / at risk) | 26/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 10 mg/kg Ipilimumab (N=40)
Cardiac arrest (Cardiac disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 3
Hyperparathyroidism (Endocrine disorders) | 1
Hypophysitis (Endocrine disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 4
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 4
Generalised oedema (General disorders) | 1
Pyrexia (General disorders) | 1
Influenza (Infections and infestations) | 1
Liver abscess (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Venous thrombosis limb (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 10 mg/kg Ipilimumab (N=40)
Tachycardia (Cardiac disorders) | 4
Adrenal insufficiency (Endocrine disorders) | 3
Hypophysitis (Endocrine disorders) | 4
Hypothyroidism (Endocrine disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 13
Constipation (Gastrointestinal disorders) | 11
Diarrhoea (Gastrointestinal disorders) | 26
Nausea (Gastrointestinal disorders) | 16
Vomiting (Gastrointestinal disorders) | 9
Chills (General disorders) | 4
Fatigue (General disorders) | 19
Pain (General disorders) | 3
Pyrexia (General disorders) | 10
Bronchitis (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 9
Alanine aminotransferase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 6
Blood alkaline phosphatase increased (Investigations) | 4
Blood creatinine increased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 8
Dehydration (Metabolism and nutrition disorders) | 11
Hyperglycaemia (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 7
Hypomagnesaemia (Metabolism and nutrition disorders) | 5
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 11
Neuropathy peripheral (Nervous system disorders) | 3
Anxiety (Psychiatric disorders) | 5
Insomnia (Psychiatric disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 3
Erythema (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 21
Rash (Skin and subcutaneous tissue disorders) | 17
Hypotension (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.